CLINICAL TRIAL: NCT00160719
Title: HLA Sensitization Following Major Cortical Allograft Bone Procedures
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 173-2005
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Bone Cancer
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: retrieve blood samples — blood samples obtain pre-op, 6 and 12 months post-op

SUMMARY:
The purpose of this study is to find out whether or not antibodies to the donor bone are present in the blood of patients who receive the donor bone.

DETAILED DESCRIPTION:
Patients who have bone cancer often have the cancerous bone removed by surgery and replaced with a piece of bone taken from a donor (a person who donates parts of their body to be used for transplants after their death). However, sometimes this replacement bone does not heal together with the patient's bone. The reason the bone does not heal is not known but it is thought that the patient's body may react to the donor bone by producing antibodies against cells on the donor bone. The purpose of this study is to find out whether or not antibodies to the donor bone are present in the blood of patients who receive the donor bone. You have been asked to participate in this study because you are scheduled to undergo this type of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients twelve years or older who are scheduled for massive fresh-frozen human structural bone allograft implantation at participating centers will be given the opportunity to participate in the study. All patients must have a reconstruction of the involved long bone with either an intercalary graft, an osteoarticular graft, or an allograft/endoprosthesis composite graft. The junction or union site studied will be the cortical-cortical, host allograft junction site, not the cancellous interfaces.

Exclusion Criteria:

* Patients who do not require major weight bearing cortical allograft bone grafts will be excluded. Also, women who are or could potentially become pregnant will be excluded from the study.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Orthopaedic clinic
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 1999-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark T. Scarborough, M.D., Principal Investigator — University of Florida
Locations (1):
- UF Orthopaedics and Sports Medicine Institute, Gainesville, Florida, United States